CLINICAL TRIAL: NCT07327229
Title: A Phase Ib/II Study of ATG-022 Plus Pembrolizumab With/Without Chemotherapy in Participants With Claudin (CLDN) 18.2-positive, HER2-negative, Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Phase Ib/II Study of ATG-022 Plus Pembrolizumab With/Without Chemotherapy in Participants With Claudin (CLDN) 18.2-positive, HER2-negative, Unresectable or Metastatic Gastric or Gastroesophageal Junction AdenocarcinomaUnresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: CLINCH-2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Antengene Biologics Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATG-022-GC-001; KEYNOTE-G37 (Other: Merck Sharp & Dohme LLC); MK-3475-G37 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2025-12-05; First posted 2026-01-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: A treatment cycle of ATG-022 will be defined as 21 days. Dosing will begin at 1.8 mg/kg Q3W with 1 subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG-022+pembrolizumab/KEYTRUDA® (Experimental)
  Interventions: Drug: ATG-022; Drug: pembrolizumab/KEYTRUDA®
- ATG-022+pembrolizumab/KEYTRUDA®+CAPOX (Active Comparator)
  Interventions: Drug: ATG-022; Drug: pembrolizumab/KEYTRUDA®; Drug: CAPOX

INTERVENTIONS:
Drug: ATG-022 — 1.8mg/kg Q3W, every 21 days as one cycle
Drug: pembrolizumab/KEYTRUDA® — 20mg Q3W, every 21 days as one cycle
Drug: CAPOX — Standard Dose level for CAPOX: Capecitabine 1000 mg/m2 PO BID on Day 1-14, Oxaliplatin 130 mg/m2 IV on Day 1, Cycled every 21 days (3 weeks) for 8 cycles.
  Arms: ATG-022+pembrolizumab/KEYTRUDA®+CAPOX

SUMMARY:
This is A Phase Ib/II Study of ATG-022 Plus Pembrolizumab With/Without Chemotherapy in Participants With Claudin (CLDN) 18.2-positive, HER2-negative, Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma

DETAILED DESCRIPTION:
This is a phase Ib/II Study of ATG-022 plus pembrolizumab with/without chemotherapy in participants with CLDN 18.2-positive, HER2-negative, PD-L1 positive (CPS≥1), unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma. Both the intervention of ATG022 + Pembrolizumab (A+P) and the intervention of ATG-022 + pembrolizumab + chemotherapy (CAPOX regimen, A+P+C) consist of a Ib and II phase.

Participants with CLDN 18.2-positive, HER2-negative, PD-L1 positive (CPS≥1) advanced or metastatic gastric or gastroesophageal junction adenocarcinoma and having progressed on or after at least one prior systemic therapy, will be enrolled in the intervention of A + P.

Participants with CLDN 18.2-positive, HER2-negative, PD-L1 positive (CPS≥1) advanced or metastatic gastric or gastroesophageal junction adenocarcinoma and having not received any prior systemic therapy, will be enrolled in the intervention of A + P + C. The study will be firstly initiated from Ib of the intervention of A+P. The initiation of the intervention of A+P+C will be based on the clinical data of A+P

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling, and analyses.
2. Aged ≥18 years as of the date of consent.
3. Histological or cytological confirmation of gastric cancer or gastroesophageal junction adenocarcinoma with CLDN 18.2 positive, HER2-negative and PD-L1 positive expression.
4. Archival tumor tissue sample within 36 months prior to participating in the study or newly obtained biopsy of a tumor lesion not previously irradiated should be provided for testing of CLDN 18.2 and PD-L1 expression for determining the criteria.
5. At least 1 measurable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 by investigators.
6. Estimated life expectancy of a minimum of 12 weeks.

Exclusion Criteria:

1. Known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during the study screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of study intervention.
2. Prior exposure to CLDN 18.2 ADC, CLDN 18.2 chimeric antigen receptor T-cell immunotherapy or agents containing MMAE.
3. Prior systemic anticancer therapy including investigational agents within 4 weeks before the first dose of study treatment or within a period during which the investigational product or systemic anticancer treatment has not been cleared from the body (e.g., a period of 5 'halflives'), whichever is the most appropriate as judged by the investigator.
4. Received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
5. Prior radiotherapy within 4 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids. Two weeks or fewer of palliative radiotherapy for non- central nervous system disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention
6. Prior a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
7. Prior major surgery (excluding placement of vascular access) within 28 days of the first dose of study treatment or minor surgical procedures≤7 days. No waiting is required following implantable port and catheter placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
AEs and SAEs | 12 months after the last subject enrolled
DLT | Up to 21 Days
  Dose Limiting Toxicity
RP2D | Up to 21 Days
  RP2D= Recommended Phase 2 Dose

SECONDARY OUTCOMES:
ORR | 12 months after the last subject enrolled
  Overall Response Rate
DOR | 12 months after the last subject enrolled
  Duration of Response
PFS | 12 months after the last subject enrolled
  Progression Free Survival
Plasma concentration of ATG-022 and derived PK paramete | One year after last patient first dose
  To characterize the PK of ATG-022

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cnacer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cnacer Hospital, Lanzhou, Gansu
  - Cancer Institute&Hospital Chinese Academy of Medical Sciences, Langfang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan Medical Hospital, Xinxiang, Henan
  - Henan Cnacer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhenghzou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Medical College of HUST, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital &Institue, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Tongren Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi provincial cancer hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of XI'AN Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical Universuty Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xiamen University, Wenzhou, Zhejiang